CLINICAL TRIAL: NCT02672592
Title: Effects of IL-1 Beta on the Hypothalamic-pituitary-gonadal (HPG) Axis in Men With Obesity and Metabolic Syndrome - The TestIL Trial
Brief Title: Effects of Interleukin-1 Beta on Low Testosterone Levels in Men With Obesity and Metabolic Syndrome
Acronym: TestIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EKNZ 2015-376
Record Dates: First submitted 2016-01-22; First posted 2016-02-03 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Hypogonadism; Metabolic Syndrome X; Obesity
Keywords: Metabolic syndrome X; Hypogonadism; Testosterone; Inflammation; Obesity
MeSH Terms: conditions — Hypogonadism; Metabolic Syndrome; Obesity; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anakinra (Active Comparator): Anakinra//Kineret® 100mg s.c. bid
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): Sodium Chloride 0.9% s.c. bid
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Anakinra — Anakinra 100mg s.c. bid
  Other Names: KINERET
  Arms: Anakinra
Drug: Sodium Chloride 0.9% — Sodium Chloride 0.9% s.c. bid
  Other Names: NaCl 0.9%
  Arms: Placebo

SUMMARY:
Obesity and the metabolic syndrome in men are associated with a high prevalence of hypogonadism of up to 50%. Increased fat mass leads to augmented release of adipocytokines and pro-inflammatory cytokines such as IL-1-beta, IL-6 and tumor necrosis factor-alpha which in turn suppress the hypothalamic-pituitary-gonadal (HPG) axis, leading to hypogonadism. This pathophysiological interplay is termed hypogonadal-obesity-adipocytokine hypothesis. TestIL is a prospective, multicenter, randomized, double-blinded, placebo-controlled trial to test the hypothesis that inhibition of IL-1-activity diminishes the inhibitory effects on HPG axis and increases testosterone levels in men with metabolic syndrome.

DETAILED DESCRIPTION:
Obesity and the metabolic syndrome are considered as chronic low-grade inflammatory states. Elevated pro-inflammatory mediators in obesity and metabolic syndrome have an inhibitory effect on the hypothalamic-pituitary-gonadal axis (HPG axis) leading to hypogonadism. Decreased testosterone production in obese men in turn promotes additional fat deposition, contributing to a vicious cycle of fat accumulation. This complex pathophysiological interplay is termed hypogonadal-obesity-adipocytokine hypothesis, describing a bidirectional relationship between low levels of testosterone and the metabolic syndrome.

TestIL is a prospective, multicenter, randomized, double-blinded, placebo-controlled trial to test the hypothesis that inhibition of IL-1-activity diminishes the inhibitory effects on HPG axis and increases testosterone levels in men with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent as documented by signature,
2. Men at the age between 18 and 75 years,
3. BMI >30 kg/m2 and at least 1 manifestation of the metabolic syndrome (i.e. prediabetes, diabetes, hypertension, dyslipidemia),
4. Total testosterone level <12 nmol/l.

Exclusion Criteria:

1. Previous or current medication with testosterone,
2. Testosterone deficiency of other cause, i.e. primary hypogonadism caused e.g. by Klinefelters syndrome, cryptorchidism, condition following orchiectomy. Known secondary hypogonadism caused by pituitary adenoma. Patients on antiandrogen medication,
3. Clinical signs of infection in the week before inclusion or history of a severe infection during the last 2 months,
4. Severe immunosuppression (e.g. patients with previously known infection with human immunodeficiency virus and a cluster of differentiation 4 (CD4) count below 350 x 109/L, patients on immunosuppressive therapy after solid organ transplantation and neutropenic patients with neutrophil count < 500 x 109/L and patients under chemotherapy with neutrophils 500-1000 x 109/L with an expected decrease to values < 500 x 109/L),
5. Hematologic disease (leukocyte count < 1.5 x 109/l, hemoglobin < 11 g/dl, platelets <100 x 103/µl),
6. Other clinically significant concomitant disease states (e.g., renal failure [Creatinine-Clearance < 30 ml/min], hepatic dysfunction [transaminases >3x upper normal range], active carcinoma,
7. History of tuberculosis,
8. Known or suspected non-compliance, drug or alcohol abuse,
9. Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to anakinra/Kineret®,
10. Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
11. Previous enrolment into the current study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Total morning testosterone (nmol/l) | 4 weeks

SECONDARY OUTCOMES:
Total morning testosterone (nmol/l) | 1 week and 3 months
Free testosterone (nmol/l) | 1 week, 4 weeks and 3 months
  Assessed by equilibrium dialysis
Bioavailable testosterone (nmol/l) | 1 week, 4 weeks and 3 months
  Assessed by equilibrium dialysis
Erectile dysfunction as assessed by International Index of Erectile Function (IIEF) score | 1 week, 4 weeks and 3 months
Clinical severity of hypogonadism as assessed by quantitative Androgen Deficiency in the Aging Male (qADAM) questionnaire | 1 week, 4 weeks and 3 months
Proportion of muscle mass as assessed by bioelectrical impedance Analysis | 1 week, 4 weeks and 3 months
Proportion of fat mass as assessed by bioelectrical impedance Analysis | 1 week, 4 weeks and 3 months
HbA1c (%) | 1 week, 4 weeks and 3 months
LH and FSH (IU/l) | 1 week, 4 weeks and 3 months
Inhibin B, ACTH (pg/ml) | 1 week, 4 weeks and 3 months
Prolactin, TSH, Insulin (mIU/l) | 1 week, 4 weeks and 3 months
Interleukin-1, Interleukin-6 (pg/ml) | 1 week, 4 weeks and 3 months
Cortisol basal (nmol/l) | 1 week, 4 weeks and 3 months
C-reactive protein (mg/l) | 1 week, 4 weeks and 3 months
free T4 (pmol/l) | 1 week, 4 weeks and 3 months
T3 (nmol/l) | 1 week, 4 weeks and 3 months
IGF-1 (nmol/l) | 1 week, 4 weeks and 3 months
GH (mU/l) | 1 week, 4 weeks and 3 months
Androstendione (μg/l) | 1 week, 4 weeks and 3 months
DHEAS (μmol/l) | 1 week, 4 weeks and 3 months
Oestradiol (pmol/l) | 1 week, 4 weeks and 3 months
Oestron (ng/l) | 1 week, 4 weeks and 3 months
17-OH-progesterone (nmol/l) | 1 week, 4 weeks and 3 months
Copeptin (pmol/l) | 1 week, 4 weeks and 3 months
Sex hormone-binding globulin (SHBG) | 1 week, 4 weeks and 3 months
Muscle strength as assessed by grip strength test | 1 week, 4 weeks and 3 months
Waist-hip-ratio | 1 week, 4 weeks and 3 months
BMI in kg/m2 | 1 week, 4 weeks and 3 months
Insulin sensitivity as assessed by homeostasis model assessment insulin resistance (HOMA-IR) | 1 week, 4 weeks and 3 months
Total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides (mmol/l) | 1 week, 4 weeks and 3 months
Leptin (μg/l) | 1 week, 4 weeks and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Professor, Principal Investigator — Endocrinology, Diabetes and Metabolism; University Hospital Basel; Beat Müller, Professor, Principal Investigator — University Department of Medicine; Kantonsspital Aarau
Locations (2):
- Switzerland (2):
  - University Department of Medicine, Kantonsspital Aarau, Aarau
  - University Hospital Basel, Basel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ebrahimi F, Urwyler SA, Betz MJ, Christ ER, Schuetz P, Mueller B, Donath MY, Christ-Crain M. Effects of interleukin-1 antagonism and corticosteroids on fibroblast growth factor-21 in patients with metabolic syndrome. Sci Rep. 2021 Apr 12;11(1):7911. doi: 10.1038/s41598-021-87207-w. PMID 33846498
- [Derived] Urwyler SA, Ebrahimi F, Burkard T, Schuetz P, Poglitsch M, Mueller B, Donath MY, Christ-Crain M. IL (Interleukin)-1 Receptor Antagonist Increases Ang (Angiotensin [1-7]) and Decreases Blood Pressure in Obese Individuals. Hypertension. 2020 Jun;75(6):1455-1463. doi: 10.1161/HYPERTENSIONAHA.119.13982. Epub 2020 Apr 10. PMID 32275191
- [Derived] Ebrahimi F, Urwyler SA, Schuetz P, Mueller B, Bernasconi L, Neyer P, Donath MY, Christ-Crain M. Effects of interleukin-1 antagonism on cortisol levels in individuals with obesity: a randomized clinical trial. Endocr Connect. 2019 Jun 1;8(6):701-708. doi: 10.1530/EC-19-0201. PMID 31042669
- [Derived] Ebrahimi F, Urwyler SA, Straumann S, Doerpfeld S, Bernasconi L, Neyer P, Schuetz P, Mueller B, Donath MY, Christ-Crain M. IL-1 Antagonism in Men With Metabolic Syndrome and Low Testosterone: A Randomized Clinical Trial. J Clin Endocrinol Metab. 2018 Sep 1;103(9):3466-3476. doi: 10.1210/jc.2018-00739. PMID 29939279